CLINICAL TRIAL: NCT03198546
Title: CAR-T Cell Targeting GPC3 for Immunotherapy of Hepatocellular Carcinoma: Phase I Clinical Trial
Brief Title: GPC3-CAR-T Cells for Immunotherapy of Cancer With GPC3 Expression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Hunan Zhaotai Yongren Medical Innovation Co. Ltd. (Other); Guangdong Zhaotai InVivo Biomedicine Co. Ltd. (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZCART-003
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma; Immunotherapy; CAR; GPC3 Gene Inactivation; T Cell; Squamous Cell Lung Cancer
Keywords: Hepatocellular carcinoma; immunotherapy; CAR-T cell therapy; GPC3 or TGFβ targeting; Phase I clinical study; squamous cell lung cancer; interventional radiology; IL7-CCL19-secreting; SCFV against PD1/CTLA4/Tigit; knockdown of PD1/HPK1; DAP10
MeSH Terms: conditions — Carcinoma, Hepatocellular; Simpson-Golabi-Behmel syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy group (Other): Appropriate patients who could benefit from the GPC3 and TGFβ targeting CAR-T cell therapy against HCC are chosen to be the CAR-T cell therapy group.
  Interventions: Biological: GPC3 and/or TGFβ targeting CAR-T cells

INTERVENTIONS:
Biological: GPC3 and/or TGFβ targeting CAR-T cells — Engineering GPC3 or/and TGFβ targeting CAR combined with/or without IL7/CCL19 and/or scfv against PD1/CTLA4/Tigit secreting vector into T cells with knockdown of PD1/HPK1, which are isolated from patients with advanced HCC, and then transfusing them back the patients.

SUMMARY:
The third/fourth generation of CAR-T cells that target GPC3 (GPC3-CART cell) and/or soluble TGFβ (GPC3/TGFβ-CART )have been constructed and their anti-HCC function has been verified by multiple in vitro and in vivo studies. Clinical studies will be performed to test the anti-cancer function by the GPC3/TGFβ-CAR-T cells in human HCC patients with GPC3 expression. In this phase I study, the safety, tolerance, and preliminary efficacy of the GPC3/TGFβ-CAR-T cell immunotherapy on human will firstly be tested.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced hepatocellular carcinoma,with written consent for this study;
2. Perform biopsy to determine the expression of GPC3 of the tumor by western blotting or IHC;
3. Collect blood from the patients and isolate mononuclear cells, activate the T cells and transfect the T cells with GPC3/TGFβ targeting CAR (or/and scfv/cytokines-secreting), amplify the number of transfected T cells as needed, test the quality and killing activity of the GPC3/TGFβ-CART cells and then transplant back the patients via systemic or local infusions (via artery or intra-tumor), and follow up closely to collect related results as needed;
4. To enhance the killing capability, CD4+ T cells are genetically engineered to express TGFβ-CAR and secret IL7/CCL19 and/or SCFVs against PD1/CTLA4/Tigit; CD8+T cells are constructed to express GPC3-DAP10-CAR with knockdown of PD1/HPK1;
5. Evaluate the clinical results as needed.
6. Will also perform the similar clinical trial on lung squamous carcinoma with the GPC3 expression.

ELIGIBILITY:
Inclusion Criteria:

1. patients with advanced HCC,which express GPC3 protein.
2. Life expectancy >12 weeks
3. Child-Pugh-Turcotte score <7
4. Adequate heart,lung,liver,kidney function
5. Available autologous transduced T cells with greater than or equal to 20% expression of GPC3 CAR determined by flow-cytometry and killing of GPC3-positive targets greater than or equal to 20% in cytotoxicity assay
6. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent. -

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Tumor size more than 25cm;
3. Severe virus infection such as HBV,HCV,HIV,et al
4. Known HIV positivity
5. History of liver transplantation
6. Active infectious disease related to bacteria, virus,fungi,et al
7. Other severe diseases that the investigators consider not appropriate;
8. Pregnant or lactating women
9. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
10. Other conditions that the investigators consider not appropriate. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | three months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GPC3-T2-CAR T cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | three months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median CAR-T cell persistence | Five years
  Median CAR-T cell persistence will be measured by quantitative rt-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jiang Z, Jiang X, Chen S, Lai Y, Wei X, Li B, Lin S, Wang S, Wu Q, Liang Q, Liu Q, Peng M, Yu F, Weng J, Du X, Pei D, Liu P, Yao Y, Xue P, Li P. Anti-GPC3-CAR T Cells Suppress the Growth of Tumor Cells in Patient-Derived Xenografts of Hepatocellular Carcinoma. Front Immunol. 2017 Jan 11;7:690. doi: 10.3389/fimmu.2016.00690. eCollection 2016. PMID 28123387
- [Derived] Pang N, Shi J, Qin L, Chen A, Tang Y, Yang H, Huang Y, Wu Q, Li X, He B, Li T, Liang B, Zhang J, Cao B, Liu M, Feng Y, Ye X, Chen X, Wang L, Tian Y, Li H, Li J, Hu H, He J, Hu Y, Zhi C, Tang Z, Gong Y, Xu F, Xu L, Fan W, Zhao M, Chen D, Lian H, Yang L, Li P, Zhang Z. IL-7 and CCL19-secreting CAR-T cell therapy for tumors with positive glypican-3 or mesothelin. J Hematol Oncol. 2021 Jul 29;14(1):118. doi: 10.1186/s13045-021-01128-9. PMID 34325726